CLINICAL TRIAL: NCT00830726
Title: Water-and Salt-homeostasis in Healthy Humans, and in Patients With Heart- or Lung Disease, Evaluated by the Excretion of Aquaporin-2 and Epithelial Sodium Channels in the Urine
Brief Title: Water- and Salt-homeostasis in Healthy Humans, and in Patients With Heart- or Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kolding Sygehus (Other)
Collaborators: Regionshospitalet Holstebro, Holstebro, Denmark (Unknown); Odense University Hospital (Other)
Responsible Party: Ole Nyvad, M.D., Kolding Hospital
Other Study IDs: S-20080141
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Healthy Volunteers; Heart Failure; Aortic Stenosis; Ischemic Heart Disease; Pulmonary Hypertension
Keywords: Aquaporin; Epithelial Sodium Channels; Heart Failure; Valvular heart disease; Ischemic heart disease
MeSH Terms: conditions — Heart Failure; Aortic Valve Stenosis; Myocardial Ischemia; Hypertension, Pulmonary; Heart Valve Diseases | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and Urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1: Healthy volunteers
- 2: Patients with symptomatic heart failure and EF < 40%
  Interventions: Drug: Pharmacologic and mechanical heart failure treatment
- 3: Patients with symptomatic aortic valve stenosis
  Interventions: Procedure: Aortic valve replacement
- 4: Patients with Acute Coronary syndromes prior to surgical intervention
  Interventions: Procedure: Revascularisation in Acute Coronary Syndrome
- 5: Patients with refractory stable angina requiring surgical intervention.
  Interventions: Procedure: Revascularisation in chronic stable angina pectoris
- 6: Patients with pulmonary hypertension and preserved systolic left ventricular function.

INTERVENTIONS:
Drug: Pharmacologic and mechanical heart failure treatment — Optimised, standard, evidence based heart failure therapy including the use of biventricular pacing.
  Groups: 2
Procedure: Aortic valve replacement — Standard aortic valve replacement as per standard criteria in the department of thoracic surgery.
  Groups: 3
Procedure: Revascularisation in Acute Coronary Syndrome — Standard percutaneous or surgical revascularisation in ACS.
  Groups: 4
Procedure: Revascularisation in chronic stable angina pectoris — Standard percutaneous or surgical revascularisation
  Groups: 5

SUMMARY:
The purpose of the study is to determine whether the excretion of renal water- and salt-channels in the urine reflects the handling of water and salt in the kidneys, and whether the excretion can be used to monitor and/or predict the effects of treatment of certain heart or lung diseases.

DETAILED DESCRIPTION:
The purpose of the study is to determine whether the excretion of renal water- and salt-channels (Aquaporin-2 and Epithelial Sodium Channels) in the urine accurately reflects the handling of water and salt in the distal tubules af the kidneys, and whether quantification of these channels in the urine is useful to monitor and/or predict the effects of pharmacologic or surgical treatment of Heart Failure and heart failure-related diseases (Aortic stenosis, acute and chronic ischemic heart disease or pulmonary hypertension)

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure
* Severe valvular aortic stenosis
* Acute Coronary Syndrome
* Medically refractory chronic angina pectoris or pulmonary hypertension with preserved left ventricular function

Exclusion Criteria:

* Pregnancy
* Drug abuse
* Malignant disease
* Significant disease of other organs including endocrine diseases

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and Outpatients and admitted patients in Kolding Hospital and Odense Universitetshospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Differences in excretion of Aquaporin-2 in urine | 6 months

SECONDARY OUTCOMES:
Differences in excretion of Epithelial Sodium Channels in urine | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ole Nyvad, M.D., Principal Investigator — Kolding Hospital, Kolding, Denmark
Locations (1):
- Kolding Hospital, Kolding, Denmark